CLINICAL TRIAL: NCT05571696
Title: Mind Matters: A High Touch, Low Cost Approach to Improving Mental Health Outcomes in Patients With Psoriatic Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elaine Husni (Other)
Collaborators: National Psoriasis Foundation (Other)
Responsible Party: Sponsor-Investigator, Elaine Husni, Staff Rheumatologist, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB#21-320
Record Dates: First submitted 2022-07-26; First posted 2022-10-07 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Arthritis, Psoriatic; Psoriasis
Keywords: Psoriatic Arthritis; Psoriasis; Mental Health; Well being
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Active Comparator): Assigned to Immune Strength program
  Interventions: Behavioral: Immune Strength
- Control Group (Active Comparator): Assigned to 12 week waitlist, receiving usual care. Study participants assigned to the wait list will receive access to Immune Strength 12 weeks after study commencement.
  Interventions: Behavioral: Immune Strength

INTERVENTIONS:
Behavioral: Immune Strength — Immune Strength is a 12 week online program that provides content, strategies, and guidance on how to improve your immune system and increase your mental wellbeing, with a focus on stress, sleep, nutrition, and exercise. In addition to the online program, each participant will be paired with a Cleveland Clinic Coach who will communicate with the participant via email. The Coach will help guide the participant throughout the program and provide encouragement and guidance for making behavior changes for making a more resilient immune system.

SUMMARY:
Despite advances in effective psoriatic disease treatment, the disease still has a serious impact on mental health and well-being of millions of patients. Up to 20.7% of patients report poor mental health, compared to 7.1% of the general population. Mental health treatment involves a combination of medication and talk therapy to address such issues. However, there is increasing evidence that optimizing behaviors such as sleep, physical activity, stress, and nutrition are critical components in improving mental health too. Numerous online health programs have evolved to help patients optimize such behaviors but very little exists for patients with psoriatic diseases. The "Immune Strength" 12 week program utilizes online electronic coaching (eCoaching) with weekly access to a wellness professional to provide a low-cost, high-touch, personalized intervention that patients can access 24/7. In conjunction with traditional clinical care, the goal of this program is to leverage the convenience, affordability, scalability and effectiveness of an online eCoaching program to improve key physical behaviors, thereby reducing the mental health burden experienced by psoriatic disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient of Cleveland Clinic
* Adults (=18 years of age)
* Diagnosis of psoriasis or psoriatic arthritis by a board certified physician.
* PHQ9 score between 5 and 20
* Computer and internet access
* A valid email address
* Able to speak & read English
* Able to understand & sign informed consent

Exclusion Criteria:

* PHQ9 score > 20
* History of major depressive disorder
* Currently receiving psychotherapy for major depressive disorder (MDD), anxiety or psychotic disorder
* On a wait-list for psychotherapeutic treatment
* Received treatment for a severe psychiatric illness in the previous 6 months
* Demonstrate a notable suicidal risk at study visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-04-14 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Patient Health Questionnaire-9 score (PHQ-9) at intervention completion. | PHQ-9 score will be collected at baseline after consent is signed and then immediately after the intervention is complete.
  The PHQ-9 is used as a screening tool for assessment of the severity of depressive symptoms.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) | PROMIS measure scores will be collected at the start of the intervention and immediately after the intervention is complete.
  PROMIS are a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Husni, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No